CLINICAL TRIAL: NCT02616341
Title: Development of a Behavioral Team Intervention for Obsessive Compulsive Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Butler Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1005-008
Record Dates: First submitted 2015-11-18; First posted 2015-11-26 (Estimated); Last update posted 2017-08-10 (Actual); Status verified 2017-08

CONDITIONS: Obsessive Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Methods; Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Team ERP (T-ERP) Intervention (Experimental): The ERP team intervention (T-ERP) consists of 25 sessions over 20 weeks with four components: (a) 3-4 pretherapy individual session with therapist, (b) 12 weekly group sessions (90-mins) led by a therapist and, (c) 10 individual coaching sessions with a case manager during weeks 2-11 of the group, and (d) 2 booster group sessions to reinforce relapse prevention
  Interventions: Behavioral: Team ERP (T-ERP) Intervention
- Treatment as Usual (TAU) (Active Comparator): Treatment as Usual (TAU) includes standard community treatment consisting of a personalized treatment plan and assistance with treatment referrals to available community resources
  Interventions: Behavioral: Treatment as Usual (TAU)

INTERVENTIONS:
Behavioral: Team ERP (T-ERP) Intervention
  Arms: Team ERP (T-ERP) Intervention
Behavioral: Treatment as Usual (TAU)
  Arms: Treatment as Usual (TAU)

SUMMARY:
The overall aim of this study is to determine modifications to Exposure and Response Prevention (ERP) therapy that are needed in order to effectively deliver treatment for Obsessive Compulsive Disorder (OCD) in a community mental health center. This study is the final study in a series of three projects executed to adapt and pilot-test a team ERP (T-ERP) intervention that will optimize therapist time by utilizing paraprofessionals to assist with group-ERP treatment plans. The intervention will be tailored to meet the unique needs of low-SES individuals with OCD and be implemented in a community mental health center (CMHC).

ELIGIBILITY:
Inclusion Criteria:

1. 18 Years to 65 Years
2. English speaking
3. Primary DSM-IV OCD (identified by the patient and therapist as the most problematic disorder over the past year)
4. At least moderate severity OCD (YBOCS > 16)
5. Not currently on psychotropic medications or on the same psychotropic medications for at least 4 weeks prior to screening
6. Have never received 10 or more sessions of ERP
7. Not currently attending psychotherapy for OCD
8. Low-income based on the U.S. Housing and Urban Development (HUDs) threshold for RI (less than $41,000 per year for individuals).

Exclusion Criteria:

1. Significant cognitive impairment (MMSE < 25)
2. Prominent suicidal ideation
3. Current psychosis, mania, alcohol or drug dependence as assessed by the SCID-P.
4. Prominent Hoarding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2012-11; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Changes in OCD symptom severity as measured by the Yale-Brown Obsessive Compulsive Scale (Y-BOCS) | Baseline, 6th week of treatment, 12th week of treatment, 3 months post-treatment, 6 months post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Maria Mancebo, Ph.D., Principal Investigator — Butler Hospital, Providence RI 02906